CLINICAL TRIAL: NCT01797380
Title: A Double-Blind, Placebo-Controlled Trial Examining the Efficacy of Escitalopram Oxalate Upon Depressive Symptoms and Fatigue in HIV Seropositive Women
Brief Title: A Trial Examining the Efficacy of Escitalopram Oxalate Upon Depressive Symptoms and Fatigue in HIV Seropositive Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00000703
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-03

CONDITIONS: Depression; HIV
Keywords: Depression; HIV
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Active Drug (Active Comparator): Escitalopram tablet, 10mg, daily, 9 weeks.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Placebo — Placebo daily for duration of double-blind portion of trial
  Arms: Sugar Pill
Drug: Escitalopram — Escitalopram 10 mg po daily for duration of double-blind portion of trial
  Arms: Active Drug

SUMMARY:
To determine the efficacy of escitalopram in treating depression in HIV seropositive women.

DETAILED DESCRIPTION:
To determine the efficacy of escitalopram in treating depression in HIV seropositive women.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression based on DSM-IV criteria;
* age 18-70 years;
* Greater than 15 on MADRS for severity of depression;
* HIV seropositive;
* no new antiviral medications over the past 2 months;
* involved in active treatment for HIV disease,
* negative serum pregnancy test
* Those subjects who are actively being treated for depression but show no improvement as defined by self-reported failure to improve with current treatment or residual depression as demonstrated by a MADRS of 15 or greater will be asked to participate in the study as well.

Exclusion Criteria:

* The presence of an active and significant psychiatric disease other than Major Depressive Disorder as diagnosed on MINI in the last 3 months;
* meeting DSM-IV criteria for an Axis I disorder within the last three months, or meeting criteria for substance abuse within the last 12 months;
* current pregnancy or lactation if breast feeding;
* history of hypersensitivity, intolerance, or contraindication to LEX;
* baseline creatinine of 2.5 or greater;
* patients taking anticoagulants;
* history of diagnosed gastric or duodenal ulcer;
* history within past year of bleeding or clotting diathesis;
* lifetime history of myocardial infarction or cerebrovascular accident;
* history of surgery within the past 3 months;
* inability to follow study procedures or complete the study;
* the use of any antidepressant medications within 5 half-lives of randomization;
* women of child-bearing potential who will not agree to use approved means of birth control during the trial;
* other reason that the primary investigator believes that the subject will be unable to complete trial or has medical/psychiatric contraindications to the trial.
* Individuals who are currently being treated for depression and show significant improvements in their depression such that discontinuing their current antidepressant therapy would likely have negative clinical consequences will be excluded from participating in this study.
* Individuals who are or become suicidal will be excluded from this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Barroso J. A review of fatigue in people with HIV infection. J Assoc Nurses AIDS Care. 1999 Sep-Oct;10(5):42-9. doi: 10.1016/S1055-3290(06)60342-7. PMID 10491802
- [Background] Currier MB, Molina G, Kato M. Citalopram treatment of major depressive disorder in Hispanic HIV and AIDS patients: a prospective study. Psychosomatics. 2004 May-Jun;45(3):210-6. doi: 10.1176/appi.psy.45.3.210. PMID 15123845
- [Background] Gutierrez MM, Rosenberg J, Abramowitz W. An evaluation of the potential for pharmacokinetic interaction between escitalopram and the cytochrome P450 3A4 inhibitor ritonavir. Clin Ther. 2003 Apr;25(4):1200-10. doi: 10.1016/s0149-2918(03)80076-0. PMID 12809966
- [Background] Himelhoch S, Medoff DR. Efficacy of antidepressant medication among HIV-positive individuals with depression: a systematic review and meta-analysis. AIDS Patient Care STDS. 2005 Dec;19(12):813-22. doi: 10.1089/apc.2005.19.813. PMID 16375613

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Active Drug
Started | 3 (Terminated due to lack of enrollment) | 2
Completed | 0 (Terminated due to lack of enrollment) | 0
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Terminated study. Study terminated prior to interventions
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Active Drug | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Depressive Symptoms
Description: Depressive symptoms were assessed by questionaire at baseline and finally at the end of the study at 9 weeks.
Time Frame: 9 weeks.
Population: Terminated due to lack of recruitment. Five subjects were consented for the trial, but were not able to complete study or generate analyzable data.
Arm/Group | Sugar Pill | Active Drug
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was terminated early due to failure to recruit.
Description: Study was terminated before adverse events were noted.No participants were treated therefore no participants were analyzed.
Arm/Group | Sugar Pill | Active Drug
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No